CLINICAL TRIAL: NCT02290249
Title: Face-to-face Intubation With Glidescope or Airtraq
Brief Title: Intubation of a Pediatric Manikin in Difficult Airway by Novice Personnel: A Comparison of Glidescope and Airtraq
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: KOU KAEK 2014/145
Record Dates: First submitted 2014-10-31; First posted 2014-11-14 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Intubation; Difficult; Edema of the Tongue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- normal airway (Active Comparator): İntubation with glidescope or airtraq in normal airway
  Interventions: Device: Glidescope; Device: Airtraq
- tongue edema (Active Comparator): intubation with glidescope or airtraq in tongue edema simulation
  Interventions: Device: Glidescope; Device: Airtraq
- face-to-face (Active Comparator): intubation with glidescope or airtraq in face-to-face intubation
  Interventions: Device: Glidescope; Device: Airtraq

INTERVENTIONS:
Device: Glidescope — Manikin was intubated by different novice personal with glidescope videolaryngoscope
Device: Airtraq — Pediatric manikin was intubated by novice personal with airtraq

SUMMARY:
Background and aims: Glidescope and Airtraq were designed to facilitate intubation and to improve teaching intubation. The investigators want to find their efficacy in normal airway, tongue edema and face-to-face orotracheal intubation models by novice personal.

Material and Methods: After Kocaeli Human Researches Ethics Committee approval, thirty six medical students who were on the beginning of their third year were enrolled in this study. After watching a video about the intubation of one of these devices, they attempted to intubate an adult manikin in three different airway models in a random order; first in normal airway, second, tongue edema and finally, in an entrapped manikin by face-to-face approach with Glidescope or Airtraq. Intubation attempts, insertion and intubation times, success rates, Cormack-Lehane grades, need of maneuvers of these devices were recorded.

DETAILED DESCRIPTION:
Trauma victims mostly had to be intubated at the scene of the area with the paramedics. In a suspect of a cervical trauma, patients must be intubated with the least movement. Videolaryngoscopic techniques had several advantages at this condition. We want to investigate which can be used easily by novice personnel.

ELIGIBILITY:
Inclusion Criteria:

* medical students at their third year,
* novice personnel

Exclusion Criteria:

* anesthesists,
* anesthesia residents,
* skilled investigators of tracheal intubation

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
intubation success rates | 5 minutes
  We recorded the first and total intubation success rates of the intubation with one of these devices

SECONDARY OUTCOMES:
intubation time | 5 minutes
  from the handling of the device till viewing the endotracheal tube entering the vocal cords
Esophageal intubation | 5 minutes
  is there an esophageal intubation occurred while inserting the tube or not
need of optimisation maneuvers | 5 minutes
  do we need an optimization maneuver while intubating or while viewing the glottis or not

CONTACTS AND LOCATIONS:
Overall Officials: Zehra I ARSLAN, Doctor, Principal Investigator — Anesthesiology and Reanimation